CLINICAL TRIAL: NCT06358729
Title: The Impact of Pre-Pregnancy Weight Loss on Infant Sucking Behavior in Response to a Challenging Nipple
Brief Title: Pre-Pregnancy Weight Loss and Baby Behavior Study
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Amanda Kinney Crandall, Research Fellow, Pediatrics, University of Michigan
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: HUM00239775
Record Dates: First submitted 2024-04-05; First posted 2024-04-11 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Obesity; Familial; Pregnancy Related; Infant Behavior
MeSH Terms: conditions — Obesity; Infant Behavior

STUDY DESIGN:
Who Masked: Participant
Masking Description: Order of nipple size use is counter-balanced, caregivers are blind to nipple size and amount of milk in the bottle (i.e., the bottle is covered) to minimize their influence over the infant's consumption. Research assistants will not be blind to nipple size as they will need to set the bottles ups for the mothers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nipple order 1 (Experimental): First the typical nipple and then challenging nipple
  Interventions: Behavioral: Typical Nipple; Behavioral: Challenging Nipple
- Nipple order 2 (Experimental): First the challenging nipple and then the typical nipple
  Interventions: Behavioral: Typical Nipple; Behavioral: Challenging Nipple

INTERVENTIONS:
Behavioral: Typical Nipple — Infants are fed their typical milk/formula by their caregiver when hungry, one feeding with their typical nipple.
Behavioral: Challenging Nipple — Infants are fed with a smaller sized nipple (i.e. with a smaller aperture, slowing the rate of milk delivery).

SUMMARY:
This study will help researchers learn more about how babies respond to bottle nipples with larger or smaller holes. Researchers guess that infants of mothers with obesity who did not lose weight prior to pregnancy will have the greatest Suck Effect on the challenging compared with the typical nipple.

DETAILED DESCRIPTION:
The researchers will recruit babies from the original cohort in the PLAN study (NCT03244722), regardless of which arms they participated in. However, the researchers will test the study arms from the original PLAN study for effects on the study's dependent variables. Their between-subjects arms included Pre-pregnancy obesity with intensive weight loss intervention, pre-pregnancy obesity with standard of care intervention, and pre-pregnancy healthy weight with no intervention. So, although the researchers are not assigning babies to any arms, their original assignment will still be assessed the study analysis.

ELIGIBILITY:
To be eligible to participate in this study...

Mother

-Current or previous participation in the PLAN study resulting in a live birth.

Child

* Mother participated in PLAN study during child's gestation
* Infant birth weight (From PLAN study records) appropriate (≥ 3rd percentile and ≤ 97th percentile) for gestational age and sex based on US Natality Data set (Oken et al, BMC Pediatrics 2003).
* Infant is 3.0 to 6.0 months old at Consent.
* Biological mother is legal guardian by maternal report.
* Biological mother is full time custodial guardian by maternal report (versus sharing custody such that infant does not live with her full time).
* Infant typically consumes at least 2 ounces in one feeding from an artificial nipple and bottle at least once per week by maternal report.
* Stated willingness by mother to comply with all study procedures and availability for the duration of the study.

Min Age: 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-02-13 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Suck effect | Up to 6 weeks
  Sucking will be measured with the NFANT® Feeding Solution

SECONDARY OUTCOMES:
Sucking pressure | Up to 6 weeks
  Sucking will be measured with the NFANT® Feeding Solution
Sucking frequency | Up to 6 weeks
  Sucking will be measured with the NFANT® Feeding Solution
Milk/Formula intake | Up to 6 weeks
Milk/Formula consumption rate | Up to 6 weeks
Number of Feedings Over 24 Hours | Up to 6 weeks
Total Hours of Sleep per 24 Hours within 24 hours of intervention | Up to 6 weeks
Total Night Wake-ups within 24 hours of intervention | Up to 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Crandall, PhD, Principal Investigator — University of Michigan; Julie Lumeng, MD, Principal Investigator — University of Michigan
Locations (1):
- The University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
The researchers may consider sharing data but hesitate due to difficulties de-identifying data of small samples. Please contact the study team if you have questions.